CLINICAL TRIAL: NCT00751088
Title: A Comparison Among Three Single-incision Devices for the Treatment of Female Urinary Genuine Stress Incontinence: a Randomized Controlled Study.
Brief Title: A Randomized Controlled Study Comparing Three Single-incision Devices for Female Urinary Stress Incontinence
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Magna Graecia (Other)
Responsible Party: Stefano Palomba, University "Magna Graecia" of Catanzaro
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 04/2008
Record Dates: First submitted 2008-09-10; First posted 2008-09-11 (Estimated); Last update posted 2013-02-27 (Estimated); Status verified 2009-07

CONDITIONS: Urinary Incontinence
Keywords: single-incision; sling; stress incontinence; surgery; treatment; Female urinary stress incontinence
MeSH Terms: conditions — Urinary Incontinence; Urinary Incontinence, Stress

ARMS (4):
- 1 (Active Comparator): Patients treated with Ajust positioning
  Interventions: Procedure: Ajust positioning
- 2 (Active Comparator): Patients treated with MiniArc positioning
  Interventions: Procedure: MiniArc positioning
- 3 (Active Comparator): Patients treated with TVT secur system
  Interventions: Procedure: TVT secur system positioning
- 4 (Active Comparator): Patients treated with tension free vaginal tape
  Interventions: Procedure: Tension free vaginal ttape

INTERVENTIONS:
Procedure: MiniArc positioning — Patient placed in lithotomic position. 1.5 cm incision made, starting 1 cm down to the urethral meatus. Tunneling wide to 12-15 mm up to the bonny edge horizontally to the inferior pubic arm by spreading the scissors blades while withdrawing it, at a plane parallel to the vaginal wall. Mucosal undermining performed at the level of the upper and lower "frenulum" attaching the sub-urethral tissue to the vaginal wall. Insertion of the device to the bonny edge, horizontaly to the inferior pubic arm, and behind the bone edge to the internal obturator muscle. MiniArc will be placed by means of curved single use needle. Incision closure.
  Arms: 2
Procedure: TVT secur system positioning — Patient placed in lithotomic position. 1.5 cm incision made, starting 1 cm down to the urethral meatus. Tunneling wide to 12-15 mm up to the bonny edge horizontally to the inferior pubic arm by spreading the scissors blades while withdrawing it, at a plane parallel to the vaginal wall. Mucosal undermining performed at the level of the upper and lower "frenulum" attaching the sub-urethral tissue to the vaginal wall. Insertion of the device to the bonny edge, horizontaly to the inferior pubic arm, and behind the bone edge to the internal obturator muscle. TVT Secur System will be placed by means of two curved, stainless steel, single use introducers. Incision closure.
  Arms: 3
Procedure: Ajust positioning — Patient placed in lithotomic position. 1.5 cm incision made, starting 1 cm down to the urethral meatus. Tunneling wide to 12-15 mm up to the bonny edge horizontally to the inferior pubic arm by spreading the scissors blades while withdrawing it, at a plane parallel to the vaginal wall. Mucosal undermining performed at the level of the upper and lower "frenulum" attaching the sub-urethral tissue to the vaginal wall. Insertion of the device to the bonny edge, horizontaly to the inferior pubic arm, and behind the bone edge to the internal obturator muscle. Ajust will be placed by means of a safe hook geometry introducer. Incision closure.
  Arms: 1
Procedure: Tension free vaginal ttape — Patient placed in lithotomic position. 15 mm vaginal incision below urethral meatus. Dissection of the paraurethral space on each side of the incision and of the bladder from the inferior edge of the pubis. Transversal 10 mm skin incisions at level of superior pubic margin. Top-down or bottom-up approach passage of the needles and sling. Adjustment of sling tension. Closure of vaginal and skin incisions.
  Arms: 4

SUMMARY:
The prevalence of urinary stress incontinence in middle age women is rated at about 30%. To date, there is an increasing use in the clinical practice of new techniques for the treatment of this condition and several surgical devices, characterized by minimally invasive approach, are commercialized.

Recently, single-incision devices have been proposed. One of the most relevant potential advantages of these devices is the possibility of performing their positioning under local anesthesia, thus, in ambulatory regimen. The employment of these devices is particularly useful in two subgroups of patients with urinary incontinence, i.e. women with genuine stress incontinence not associated to pelvic organ prolapse (POP) and women whose stress incontinence raised after surgical correction of (severe) POP.

Poor data coming from randomized controlled trials (RCTs) are available regarding single-incision devices for the treatment of stress incontinence, and there are no conclusions in terms of their feasibility, efficacy and safety. Finally, to our knowledge no randomized controlled trial is actually available in literature comparing different single-incision devices.

DETAILED DESCRIPTION:
Women with genuine urinary stress incontinence not associated with POP will be enrolled and randomized in three groups (arm 1, arm 2 and arm 3). All patients eligible will undergo baseline assessment consisting of anthropometric, clinical, hormonal, ultrasonographic and urodynamic evaluations. At time of surgery, all patients will be randomized in three surgical treatment groups (arm 1, 2 and 3). Patients of arm 1 will be treated with positioning of Ajust (Bard Urological Division, Covington, GA, USA), patients of group 2 will be treated with positioning of MiniArc (AMS, Minnetonka, MN, USA) and patients of arm 3 will be treated with positioning of TVT Secur System (Ethicon, Somerville, NJ, USA).

During the study, the clinical outcomes, and the adverse experience will be evaluated in each patient.

Data will be analyzed using the intention-to-treat principle and a P value of 0.05 or less will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* genuine stress incontinence

Exclusion Criteria:

* pregnancy
* <12 months postpartum
* systemic disease and/or drugs known to affect bladder function
* current chemotherapy or radiation therapy
* urethral diverticulum
* augmentation cytoplasty
* artificial sphincter
* genital prolapse equal to or more than second degree
* history of severe abdominopelvic infections
* detrusor instability and/or intrinsic sphincter dysfunction
* other gynecologic pathologies
* BMI >30

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2008-09

PRIMARY OUTCOMES:
Subjective cure rate (compared to results of TVT)

SECONDARY OUTCOMES:
Objective cure rate
Intraoperative complication rate | one day
Blood loss
Postoperative complication rate | thirty days
Long-term complication rate | twelve months
Postoperative pain
Patients' satisfaction
Sexual function
Quality of life
Recurrence rate
Feasibility (degree of surgical difficulty in non-trained surgeons)
Learning curve (change in operative time, intra- and post-operative complications over the time

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Palomba, MD, Principal Investigator — Chair of Obstetrics and Gynecology, University "Magna Graecia" of Catanzaro; Fulvio Zullo, MD, Study Chair — Chair of Obstetrics and Gynecology, University "Magna Graecia" of Catanzaro
Locations (1):
- "Pugliese" Hospital, Catanzaro, Catanzaro, Italy

REFERENCES:
- [Derived] Carter E, Johnson EE, Still M, Al-Assaf AS, Bryant A, Aluko P, Jeffery ST, Nambiar A. Single-incision sling operations for urinary incontinence in women. Cochrane Database Syst Rev. 2023 Oct 27;10(10):CD008709. doi: 10.1002/14651858.CD008709.pub4. PMID 37888839
- [Derived] Palomba S, Falbo A, Oppedisano R, Torella M, Materazzo C, Maiorana A, Tolino A, Mastrantonio P, La Sala GB, Alio L, Colacurci N, Zullo F; SIMS Italian Group. A randomized controlled trial comparing three single-incision minislings for stress urinary incontinence. Int Urogynecol J. 2014 Oct;25(10):1333-41. doi: 10.1007/s00192-014-2383-0. Epub 2014 Apr 16. PMID 24737301
- [Derived] Palomba S, Oppedisano R, Falbo A, Torella M, Maiorana A, Materazzo C, Tolino A, Mastrantonio P, La Sala GB, Alio L, Colacurci N, Zullo F; SIMS Italian Group. Single-incision mini-slings versus retropubic tension-free vaginal tapes: a multicenter clinical trial. J Minim Invasive Gynecol. 2014 Mar-Apr;21(2):303-10. doi: 10.1016/j.jmig.2013.08.714. Epub 2013 Oct 19. PMID 24148568
- [Derived] Palomba S, Oppedisano R, Torella M, Falbo A, Maiorana A, Materazzo C, Tartaglia E, Tolino A, Mastrantonio P, Alio L, Colacurci N, Zullo F; SIMS Italian Group. A randomized controlled trial comparing three vaginal kits of single-incision mini-slings for stress urinary incontinence: surgical data. Eur J Obstet Gynecol Reprod Biol. 2012 Jul;163(1):108-12. doi: 10.1016/j.ejogrb.2012.03.038. Epub 2012 May 1. PMID 22552180